CLINICAL TRIAL: NCT02810860
Title: A Study to Pilot the Use of a Multimedia Application to Collect the Largest PROMs (Patient Reported Outcome Measures) Dataset in Adult Patients Undergoing Elective Laparoscopic Cholecystectomy for Symptomatic Gallstones and to Aid the Informed Consent Process
Brief Title: Multimedia Informed Consent & PROMs in Laparoscopic Cholecystectomy
Acronym: EPICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: EIDO Healthcare (Other); The Royal College of Surgeons of England (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15GS002
Record Dates: First submitted 2016-04-25; First posted 2016-06-23 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2016-12

CONDITIONS: Gallstone Disease
Keywords: laparoscopic cholecystectomy
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Other): Administration of a disease-specific and generic PROMs survey to patients undergoing Laparoscopic Cholecystectomy
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Administration of a disease-specific and generic PROMs survey to patients undergoing Laparoscopic Cholecystectomy

SUMMARY:
Collection of PROMs (Patient Reported Outcome Measures) data from patients before and after an operation to remove their gallbladder for the treatment of symptomatic gallstones. This PROMs data will provide information to clinicians and trusts about the health gain following this type of surgery and the impact on patient's quality of life.

This information will be collected by the implementation of the patient Website aboutmyop.org. This will not only allow patients to complete quality of life (PROMs) questionnaires online, but will also allow them to access information on their condition and necessary surgery, in addition to post-operative follow-up.

DETAILED DESCRIPTION:
Patients referred with gallstone disease necessitating surgery (laparoscopic cholecystectomy) will be invited to engage with our on-line interactive website. This will allow a two-way exchange of information in a secure environment (N3 compliant) to inform the patient about the risks, benefits, alternatives to surgery (cholecystectomy), and post- operative expectations. Furthermore, it will inform clinicians about the patient's symptoms and history, and record a pre-operative Patient Reported Outcome Measure (PROM). The patient's understanding of the facts required for informed consent will be measured and a "Patient Health & Understanding Report" generated for hospital clinicians. This will form part of the electronic patient record, and will be a medico-legal document.

As with current practice patients will still attend their initial outpatient clinic appointment where they will meet a surgeon who will determine the appropriateness of surgery. Informed consent for surgery (cholecystectomy) will be obtained at this initial consultation facilitated by the information obtained from the "Patient Health & Understanding Report". The patient will then continue to interact with the on-line platform before and after their operation to ensure they are well informed and to monitor their post-operative progress.

7 days after surgery the patient will be prompted to interact with the website to answer questions about their progress and recovery. This will replace the existing telephone follow-up interaction. Any problems identified will trigger a protocol driven interaction between the hospital and the patient.

At 1, 3 and 6 months after surgery a post-operative PROMs questionnaire will be answered by the patient allowing comparison of pre- and post-operative PROMs. This study will lead to the largest PROMs assessment of the effectiveness of laparoscopic cholecystectomy, will study the feasibility of our Website as a multimedia application in assisting with the process of informed consent, and will determine whether telephone follow-up can be safely replaced by a protocol driven online system.

ELIGIBILITY:
Inclusion Criteria:

Male or female.

* Adults:aged 18 to 85 years.
* Be referred for consideration for an elective laparoscopic cholecystectomy for symptomatic gallstones based on their GPs diagnosis and referral to a general surgeon.
* Patients initially listed for laparoscopic cholecystectomy but subsequently converted to open cholecystectomy or subsequently have a more complex 'biliary' procedure (including but not exclusive to bile duct exploration, biliary drain insertion, biliary bypass procedure).

Exclusion Criteria:

* Patients unable to, or those choosing not to engage with the multimedia process --- including patients lacking mental capacity, patients who do not have access to a multimedia device (including but not exclusive to a computer, tablet or multimedia phone), patients who are unable to use a multimedia device unassisted.
* Patients who are unable to read or communicate n English without the presence of a translator.
* Patients undergoing another major non---biliary operation during the same operation as their cholecystectomy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Mean domain PROMs scores for each study participant | 30-Days,3 Months and 6 Months
  We will look at the change in score between: pre--op and 30-Days, Pre-op and 3 Months post-op and pre-op and 6 months post-op. For this analysis we hope to use the paired t---test, however depending on whether the data is normally distributed or not this may require non---parametric analyses with the Wilcoxon rank---sum test. We also aim to look at the overall trend, which will require analysis of variance.

SECONDARY OUTCOMES:
Completion of the Multimedia Informed Consent package on aboutmyop.org | 30 days
Completion of the 7---Day follow---up questionnaire. | 7 days
Completion of a Patient Satisfaction Survey to receive feedback on the process. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prita Daliya, MBChB, MRCS, PGDip(Hons), Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daliya P, Carvell J, Rozentals J, Lobo DN, Parsons SL. Digital Follow-Up After Elective Laparoscopic Cholecystectomy: A Feasibility Study. World J Surg. 2022 Nov;46(11):2648-2658. doi: 10.1007/s00268-022-06684-w. Epub 2022 Aug 11. PMID 35953737